CLINICAL TRIAL: NCT03874221
Title: Automatic Retinal Image Analysis (ARIA) to Predict Coronary Artery Disease in HIV-infected Individuals
Brief Title: ARIA to Predict Coronary Artery Disease in HIV-infected Individuals
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: ARIA protocol v.1. 21012019
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hiv; Coronary Artery Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — : Peripheral blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With effective anti-retroviral therapy, non-communicable diseases, such as cardiovascular diseases, have become the major cause of morbidity and mortality for people living with HIV. There is only limited data evaluating the burden and risk factors of cardiovascular disease in the Asian HIV-infected population. Accurate non-invasive tools for prediction of cardiovascular disease, particularly in Asian HIV-infected populations, are urgently needed. Recently, more detailed evaluation of the complex retinal vasculature has been made feasible with advances in digitalized retinal imaging techniques.

This study aims 1. to determine the prevalence of coronary atherosclerosis and obstructive coronary artery disease HIV-infected individuals with one or more cardiovascular disease risk factors in Asia. 2. to determine the performance of automatic retinal image analysis (ARIA) in predicting the risk of coronary artery disease in HIV-infected individuals, as compared to traditional risk prediction tools. Patients will undergo a coronary CT angiogram, followed by an automatic retinal image analysis within 4 weeks post completion of CT angiogram.

ELIGIBILITY:
Inclusion Criteria:

* Positive anti-HIV antibody
* Age 30 or above
* Presence of one or more risk factors for cardiovascular disease

Exclusion Criteria:

* Presence of overt coronary artery disease
* Impaired renal function
* Allergy to intravenous contrast
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HIV-infected individuals followed up in Metabolic Research Clinic and Infectious Diseases clinic of the Prince of Wales Hospital will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Coronary atherosclerosis defined as the presence of any plaque in one or more coronary artery segments | 1 year

SECONDARY OUTCOMES:
Presence of any CAC, Presence of significant CAC, Obstructive coronary artery disease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lui, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No